CLINICAL TRIAL: NCT01606059
Title: A Randomized, Open Label, 2-treatment, 2-sequence, Cross-over Study to Compare the Safety and Pharmacokinetics of DW-0919 and DW-0920 After Single Oral Administration in Healthy Male Volunteers
Brief Title: Phase 1 Study of DW-0919 & DW-0920 in Healthy Male Volunteers Under Fasting Condition
Acronym: DW0919-1003
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Collaborators: Chungnam National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: DW0919-1003
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
MeSH Terms: interventions — Acetaminophen; Tramadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DW-0919 (Active Comparator)
  Interventions: Drug: DW-0919
- DW-0920 (Experimental)
  Interventions: Drug: DW-0920

INTERVENTIONS:
Drug: DW-0920 — Dosage form: Extended release tablet Dosage: 2 tablets
  Other Names: Acetaminophen: 325mg; Tramadol: 37.5mg; Wontran ER tab.
  Arms: DW-0920
Drug: DW-0919 — Dosage form: Extended release tablet Dosage: 1 tablet
  Other Names: Acetaminophen: 650mg; Tramadol: 75mg
  Arms: DW-0919

SUMMARY:
The purpose of this study is to evaluate safety and pharmacokinetics of DW-0919 and DW-0920 in healthy male volunteers under fasting condition.

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 20 to 55 years at screening.
* No significant congenital/chronic disease.
* No symptoms in physical examination.
* Appropriate subjects as determined by past medical history, laboratory tests, serology and urinalysis.
* Be able to understand the objective, method of the study, the characteristics of investigational drug, and comply with the requirement of the study. Subject must provide written informed consent prior to study participation.

Exclusion Criteria:

* History of Hyperreactivity with drug ingredients(acetaminophen, tramadol) or opioids.
* History or presence of liver, kidney, or nervous system disease, respiratory disorders, endocrinological disorders, hemato-oncologic, cardiovascular or psychiatric or cognitive disorders.
* History of gastrointestinal disorders (bleeding, ulceration, hemorrhoids, piles) or disorders of absorption, distribution, metabolism, excretion.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
AUC of DW-0919(Acetaminophen, Tramadol) | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36
Cmax of DW-0919(Acetaminophen, Tramadol) | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36
AUC of DW-0920(Acetaminophen, Tramadol) | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36
Cmax of DW-0920(Acetaminophen, Tramadol) | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

REFERENCES:
- [Derived] Kim HC, Yoon DY, Lee S, Jang IJ, Hong JH, Kim J. Comparative pharmacokinetics between two tablets of tramadol 37.5 mg/acetaminophen 325 mg and one tablet of tramadol 75 mg/acetaminophen 650 mg for extended-release fixed-dose combination. Transl Clin Pharmacol. 2022 Jun;30(2):112-119. doi: 10.12793/tcp.2022.30.e12. Epub 2022 Jun 27. PMID 35800670